CLINICAL TRIAL: NCT04229498
Title: Comparison of Clinical Outcomes in Bloodstream Infections With Carbapenem Hetero-resistant vs Carbapenem Resistant Klebsiella Pneumoniae (COMBAT)
Brief Title: Comparison of Bloodstream Infections With Carbapenem Hetero-resistant vs Carbapenem Resistant Klebsiella Pneumoniae
Acronym: COMBAT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: SCARE (Study group for carbapenem resistance) (Other)
Responsible Party: Sponsor
Other Study IDs: COMBAT121219
Record Dates: First submitted 2020-01-04; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Bloodstream Infection
Keywords: Carbapenem resistant Klebsiella pneumoniae; Carbapenem heteroresistant Klebsiella pneumoniae; Bloodstream Infections; Sepsis; Septic shock; Relapses/re-infections; Mortality
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Combined Modality Therapy; Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood culture samples of participants
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Carbapenem resistant Klebsiella pneumoniae group: Participants having bloodstream infection caused by carbapenem-resistant Klebsiella pneumoniae and systemic signs of infection. Only first bloodstream infection episode will be included for each participant
  Interventions: Drug: Monotherapy and combination therapy (all antibiotics that are given by attending pysicians and can be active against Klebsiella pneumoniae will be evaluated)
- Carbapenem hetero-resistant Klebsiella pneumoniae group: Participants having bloodstream infection caused by carbapenem-heteroresistant Klebsiella pneumoniae and systemic signs of infection. Only first bloodstream infection episode will be included for each participant
  Interventions: Drug: Monotherapy and combination therapy (all antibiotics that are given by attending pysicians and can be active against Klebsiella pneumoniae will be evaluated)

INTERVENTIONS:
Drug: Monotherapy and combination therapy (all antibiotics that are given by attending pysicians and can be active against Klebsiella pneumoniae will be evaluated) — In carbapenem heteroresistant Klebsiella pneumoniae group, carbapenem monotherapy (ertapenem, imipenem, meropenem) vs other treatment groups will also be compared
  Other Names: Drug

SUMMARY:
COMBAT trial was contemplated to elucidate unknown clinical relevance of carbapenem heteroresistance among Klebsiella pneumoniae species. Bloodstream infections, type of frequently seen invasive infections that pathogen isolation, identification of antimicrobial resistance mechanisms can be performed efficiently, with carbapenem resistant Klebsiella pneumoniae (CRKp) and carbapenem hetero-resistant Klebsiella pneumoniae will be compared in terms of relevant clinical outcomes such as 30-day mortality rate, 14-day clinical cure rate, 7-day microbiological eradication rate and 90-day relapse/re-infection rate. In addition, underlying molecular resistance mechanisms causing carbapenem hetero-resistance among Klebsiella pneumoniae isolates will be investigated by using whole genome sequences.

DETAILED DESCRIPTION:
Main Objectives:

1. Conceiving the clinical relevance of carbapenem hetero-resistance phenomenon among Klebsiella pneumoniae strains.
2. Identification of molecular resistance mechanisms causing carbapenem hetero-resistance among Klebsiella pneumoniae strains
3. Identification of accuracy of gradient test (e.g. E-test) and disc diffusion test for detection of carbapenem heteroresistance as compared with gold standard PAP analysis

Hypothesis

Main hypothesis

1- 30-day mortality rate is higher in bloodstream infections caused by CRKp than carbapenem hetero-resistant Klebsiella pneumoniae

Secondary hypothesis

1. 90-day relapse/re-infection rates are similar in CRKp and carbapenem heteroresistant Kp groups. However, carbapenem monotherapy is associated with higher rate of relapse/reinfection rate in treatment of bloodstream infection caused by carbapenem heteoresistant K. pneumonia even if used as high dose and prolonged infusion regimens.
2. 14-day clinical cure rate is significantly higher in carbapenem heteroresistant Kp group than CRKp group.
3. 14-day clinical cure rate is significantly lower in patients having BSI caused by carbapenem hetero-resistant K. pneumoniae and treated with carbapenem monotherapy.
4. 7-day microbiological cure rate is significantly higher in carbapenem heteroresistant Kp group than CRKp group.
5. 7-day microbiological cure rate is significantly lower in patients having BSI caused by carbapenem heteroresistant K. pneumoniae and treated with carbapenem monotherapy.

Study Design:

Prospective multi-centre multinational study

Setting and study period:

Tertiary care hospitals form different parts of the world will be included in COMBAT trial. Study period is scheduled to be 01.04.2020-01.04.2021 or longer until pre-defined sample size is attained. Local (primary) investigators will collect microbiological and clinical data of participants. Site investigators will screen the microbiology laboratory data in daily interval to identify patients with CRKp or carbapenem hetero-resistant Kp bacteremia. All consecutive patients with monobacterial CRKp or carbapenem hetero-resistant Kp BSI will be eligible to be evaluated for inclusion in the study. Carbapenem resistance will be determined according to 2015 CDC criteria. The presence of carbapenem hetero-resistance among Kp blood culture isolates will be initially determined based on observation of some sub-colonies in inhibition zone of carbapenems. The presence of hetero-resistance against only one type of carbapenems including ertapenem, imipenem, meroepenem will be sufficient to be included. Identification of carbapenem hetero-resistant subpopulations is not infrequent while performing disc diffusion tests or gradient tests (eg. E-test) in our daily practices. However, the exact sensitivity and specificity of these tests for identification of carbapenem hetero-resistance among gram-negative microorganisms are not known yet. The participants with BSI caused by carbapenem hetero-resistant Kp that is defined by disc diffusion or gradient test results will be recruited into carbapenem hetero-resistant Kp group. However, clinical carbapenem hetero-resistant Kp isolates will be transfered to pre-defined reference centres of each country via appropriate transfer culture media. Population analysis profiling (PAP) will be performed for these pathogens in reference centres. Although PAP is recommended method for identification of carbapenem hetero-resistance, it is cumbersome for microbiology laboratories for routine usage. Participants suspected of having BSI with carbapenem hetero-resistant Kp based on routine microbiological methods will be initially included and data of these patients will be recorded but, these patients will be excluded from our final analysis if PAP analysis does not confirm the presence of carbapenem hetero-resistance in these pathogens. PAP analysis will be used as a confirmatory test for identification of carbapenem heteroresistance among Klebsiella pneumoniae isolates. PAP will be performed at the end of patient recruitment and after collection of all isolates in reference centers. Therefore, treatment decisions and any other interventions will not be affected by the results of PAP analysis. PAP will only be used for identification of presence of carbapenem hetero-resistance among suspicious isolates as a gold standard method. This study will be purely observational and no intervention will be in any part of patient follow-up (eg. diagnosis, treatment etc.) and all decisions will be taken by attending physicians. Briefly, PAP analysis will be performed as following: one colony from a culture grown overnight on Columbia agar is inoculated into 5 ml of Luria-Bertani broth. After 24 h of incubation, 0.1 ml of bacterial suspension with a density corresponding 0.5 McFarland is serially diluted and spread onto Mueller-Hinton agar containing two-fold serial dilutions of meropenem, imipenem, ertapenem with concentrations ranging from 0.25 to 256 mg/L. One hundred microliters of ten-fold serial dilution(s) of a 0.5 McFarland suspension is spread on drug-free Mueller-Hinton agar and incubated for 48h at 37 °C to determine the CFUs/ml. Colony counts from three replicate plates are performed for all of the isolates, and mean values are estimated. The number of resistant cells in 0.1 ml of starting bacterial suspension is calculated and the log CFUs/ml is plotted against the antibiotic concentration. The frequency of hetero-resistant subpopulations at the highest drug concentration will be calculated and divided the number of colonies grown on antibiotic-containing plates by the colony counts from the same bacterial inoculum plated onto antibiotic-free plates. A protocol for PAP analysis will be prepared and send to reference centers to perform PAP more smoothly and with same techniques in each reference centers. Site investigators will also collect CRKp isolates and keep these isolates in appropriate conditions until time of transfer for analysis. All CRKp isolates will be sent to the central microbiology laboratories in each country for identification of carbapenemase genes by performing multiplex PCR (polymerized chain reaction).

Sample Size:

To best of our knowledge, there is no study investigating clinical outcomes of bloodstream or other type of invasive infections caused by carbapenem hetero-resistant gram negative bacteria in literature. Therefore, this study will be conducted as a pilot study. Nevertheless, 200 participants for CRKp arm and 100 participants for carbapenem hetero-resistant Klebsiella pneumonaie arm are planned to be involved.

Follow-up:

Participants will be evaluated for microbiological eradication on day 7 by control blood cultures and cultures of primary infection source. If causative pathogen is not eradicated within 7 days follow-up, consecutive cultures will be taken between 7-28 days as being necessary. Patients will also be evaluated for clinical response on day-7 and day-14 by using relevant parameters. All participants will be followed for 90 days after index blood culture date. During this follow-up period, regular assessment starting from blood culture sampling will be carried out and participants will be primarily evaluated for occurrence of any infection (blood stream or other type of invasive infection) in once a month interval if the participants are discharged. Participants will be warned to apply to our centres until the completion of 90-day follow-up period when symptoms of infection develop (eg fever, chills). Also, participants will be informed to call physicians who are primary investigators of particular centre in this study when the participants arrive to hospital clinic or emergency department. Primary investigators will evaluate participants and send their culture samples according to clinical necessity. After review of the results of cultures and clinical presentation, the patients will be allocated into infections with carbapenem resistant or carbapenem hetero-resistant Klebsiella pneumoniae groups. If the participant is discharged before completion of the 90-days, he/she will be contacted in 30 days interval by telephone call to appraise the investigated outcomes.

Microbiological Analysis:

* Antimicrobial susceptibility tests (AST) will be performed in each center and not be repeated. Therefore, AST results will be obtained from hospital database.
* PAP (Population analysis profiling) will be performed in reference centers in each country to identify actual hetero-resistant isolates among suspected isolates in which some subpopulations within inhibition zone in gradient test (eg.E-test) or disk diffusion test are identified
* Multiplex PCR will be used for identification of types of carbapenemase (will be performed in reference centers)
* Whole genome sequencing will be used to identifiy molecular mechanisms of carbapenem hetero-resistance in clinical isolates (will be performed in reference centers)
* Colistin resistance will be investigated by broth microdilution method (will be performed in reference centers)
* EUCAST breakpoints will be used for identification of resistance against all antibiotics except tigecycline in which FDA breakpoints will be applied.
* The results of antimicrobial susceptiblity and MIC values of carbapenems, colistin, tigecycline, amikacin and gentamycin will be indicated for most resistant subpopulations identified in PAP analysis. MIC values of aforementioned antibiotics will be analyzed in reference centers by using broth microdilution method. For other antibiotics, AST results of parental isolates will be recorded and obtained from hospital database.

Statistical Analysis:

Variables were described using median (interquartile range) or frequency count according to the type of variable. The categorical variables will be compared by Pearson's chi-square or Fisher's exact test if cells have a frequency of 5 or less and continuous variables by Wilcoxon-Mann-Whitney U tests for nonnormally distributed variables or Student's t test for normally distributed variables. The groups (CRKp vs Carbapenem hetero-resisant) were compared by using univariate analysis to define the variables that have significant difference between comparison groups. All univariables with a P value of 0.20 or less will be included in the multivariate Cox regression models by manually selecting them in a backward stepwise manner according to clinical value and their association. VIF (variance inflation factor) will be calculated for each variables incorporated into multivariate model. The best fit model will be picked up according to likelihood ratio test. In another analysis comparing CRKp group and carbapenem hetero-resistant group, a propensity score will be calculated and this score will be incorporated into cox regression analysis model as a confounding parameter. Cox reggression analysis will be applied to compare relevant outcomes such as 30-day mortality and 14-day clinical cure rates.

Survival for 30 days from the first positive blood culture was plotted as Kaplan-Meier curves and the rates of survival were compared by the log rank test to evaluate the effect of carbapenem hetero-resistance. All tests were two-tailed, and significance was set at 0.05 in SPSS software (version 20.0; SPSS Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* All adult (≥18 years) patients who have monobacterial BSI with CRKp or carbapenem hetero-resistant Klebsiella pneumoniae except palliative patients and pregnant or breast-feeding patients

Exclusion Criteria:

* • <18 years old patients

  * Palliative patients
  * Pregnant or breast-feeding patients
  * Subsequent BSI episodes in the same patients (only first episode will be included)
  * Polimicrobial bacteremia
  * Patients who are not followed and treated by infectious diseases physicians
  * Patients who die within 24 hours after onset of BSI which is defined as the time in which the sample for blood culture is taken.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (≥18 years) patients who have monobacterial BSI with CRKp or carbapenem hetero-resistant Klebsiella pneumoniae and treated by infectious diseases specialist will be inculded except palliative patients and pregnant or breast-feeding patients. Participants having polimicrobial BSI episode (more than 1 microorganism identified in blood culture) and subsequent BSI episodes caused by CRKp or carbapenem heteroresistant Klebsiella pneumoniae will be excluded.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
30-day crude mortality | 30-day
  Death by any cause

SECONDARY OUTCOMES:
14-day clinical response | 14-days
  Complete response: Improvement in clinical response resulting in ceasing of antibiotic therapy.
  Partial response: Improvement in clinical response with continuation of antibiotic therapy.
  No response: No improvement
90-day relapse or re-infection | 90-days
  Relapse/Re-infection: Any type of invasive infections including BSI caused by carbapenem resistant or carbapenem hetero-resistant Kp within 90 days of index BSI

OTHER OUTCOMES:
7-day microbiological eradication | 7-day
  No growth in follow-up culture taken within 7 days of index blood culture
Resistance genes | 90 days
  Whole genome sequences will be used to identify genetic mechanisms (presumably causative genes) of carbapenem hetero-resistance among Klebsiella pneumoniae clinical isolates

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah T Aslan, Dr., Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Any data will not be shared with other researchers except the data of participants recruited from their centers.

REFERENCES:
- [Background] Alexander HE, Leidy G. MODE OF ACTION OF STREPTOMYCIN ON TYPE b HEMOPHILUS INFLUENZAE : II. NATURE OF RESISTANT VARIANTS. J Exp Med. 1947 May 31;85(6):607-21. doi: 10.1084/jem.85.6.607. PMID 19871639
- [Background] SUTHERLAND R, ROLINSON GN. CHARACTERISTICS OF METHICILLIN-RESISTANT STAPHYLOCOCCI. J Bacteriol. 1964 Apr;87(4):887-99. doi: 10.1128/jb.87.4.887-899.1964. PMID 14137628
- [Background] Kayser FH, Benner EJ, Hoeprich PD. Acquired and native resistance of Staphylococcus aureus to cephalexin and other beta-lactam antibiotics. Appl Microbiol. 1970 Jul;20(1):1-5. doi: 10.1128/am.20.1.1-5.1970. PMID 5201887
- [Background] Wright GD, Sutherland AD. New strategies for combating multidrug-resistant bacteria. Trends Mol Med. 2007 Jun;13(6):260-7. doi: 10.1016/j.molmed.2007.04.004. Epub 2007 May 9. PMID 17493872
- [Background] El-Halfawy OM, Valvano MA. Chemical communication of antibiotic resistance by a highly resistant subpopulation of bacterial cells. PLoS One. 2013 Jul 3;8(7):e68874. doi: 10.1371/journal.pone.0068874. Print 2013. PMID 23844246
- [Background] Ryffel C, Strassle A, Kayser FH, Berger-Bachi B. Mechanisms of heteroresistance in methicillin-resistant Staphylococcus aureus. Antimicrob Agents Chemother. 1994 Apr;38(4):724-8. doi: 10.1128/AAC.38.4.724. PMID 8031036
- [Background] Hallander HO, Laurell G. Identification of cephalosporin-resistant Staphylococcus aureus with the disc diffusion method. Antimicrob Agents Chemother. 1972 May;1(5):422-6. doi: 10.1128/AAC.1.5.422. PMID 4670484
- [Background] Kondo N, Kuwahara-Arai K, Kuroda-Murakami H, Tateda-Suzuki E, Hiramatsu K. Eagle-type methicillin resistance: new phenotype of high methicillin resistance under mec regulator gene control. Antimicrob Agents Chemother. 2001 Mar;45(3):815-24. doi: 10.1128/AAC.45.3.815-824.2001. PMID 11181367
- [Background] Khosrovaneh A, Riederer K, Saeed S, Tabriz MS, Shah AR, Hanna MM, Sharma M, Johnson LB, Fakih MG, Khatib R. Frequency of reduced vancomycin susceptibility and heterogeneous subpopulation in persistent or recurrent methicillin-resistant Staphylococcus aureus bacteremia. Clin Infect Dis. 2004 May 1;38(9):1328-30. doi: 10.1086/383036. Epub 2004 Apr 14. PMID 15127350
- [Background] Park KH, Kim ES, Kim HS, Park SJ, Bang KM, Park HJ, Park SY, Moon SM, Chong YP, Kim SH, Lee SO, Choi SH, Jeong JY, Kim MN, Woo JH, Kim YS. Comparison of the clinical features, bacterial genotypes and outcomes of patients with bacteraemia due to heteroresistant vancomycin-intermediate Staphylococcus aureus and vancomycin-susceptible S. aureus. J Antimicrob Chemother. 2012 Aug;67(8):1843-9. doi: 10.1093/jac/dks131. Epub 2012 Apr 25. PMID 22535621
- [Background] Rodriguez CH, Bombicino K, Granados G, Nastro M, Vay C, Famiglietti A. Selection of colistin-resistant Acinetobacter baumannii isolates in postneurosurgical meningitis in an intensive care unit with high presence of heteroresistance to colistin. Diagn Microbiol Infect Dis. 2009 Oct;65(2):188-91. doi: 10.1016/j.diagmicrobio.2009.05.019. PMID 19748431
- [Background] Charles PG, Ward PB, Johnson PD, Howden BP, Grayson ML. Clinical features associated with bacteremia due to heterogeneous vancomycin-intermediate Staphylococcus aureus. Clin Infect Dis. 2004 Feb 1;38(3):448-51. doi: 10.1086/381093. Epub 2004 Jan 12. PMID 14727222
- [Background] Weel JF, van der Hulst RW, Gerrits Y, Tytgat GN, van der Ende A, Dankert J. Heterogeneity in susceptibility to metronidazole among Helicobacter pylori isolates from patients with gastritis or peptic ulcer disease. J Clin Microbiol. 1996 Sep;34(9):2158-62. doi: 10.1128/jcm.34.9.2158-2162.1996. PMID 8862577
- [Background] Fusco DN, Alexander EL, Weisenberg SA, Mediavilla JR, Kreiswirth BN, Schuetz AN, Jenkins SG, Rhee KY. Clinical failure of vancomycin in a dialysis patient with methicillin-susceptible vancomycin-heteroresistant S. aureus. Diagn Microbiol Infect Dis. 2009 Oct;65(2):180-3. doi: 10.1016/j.diagmicrobio.2009.05.017. PMID 19748429
- [Background] van Hal SJ, Jones M, Gosbell IB, Paterson DL. Vancomycin heteroresistance is associated with reduced mortality in ST239 methicillin-resistant Staphylococcus aureus blood stream infections. PLoS One. 2011;6(6):e21217. doi: 10.1371/journal.pone.0021217. Epub 2011 Jun 21. PMID 21713004
- [Background] Sola C, Lamberghini RO, Ciarlantini M, Egea AL, Gonzalez P, Diaz EG, Huerta V, Gonzalez J, Corso A, Vilaro M, Petiti JP, Torres A, Vindel A, Bocco JL. Heterogeneous vancomycin-intermediate susceptibility in a community-associated methicillin-resistant Staphylococcus aureus epidemic clone, in a case of Infective Endocarditis in Argentina. Ann Clin Microbiol Antimicrob. 2011 Apr 28;10:15. doi: 10.1186/1476-0711-10-15. PMID 21527033
- [Background] Campanile F, Bongiorno D, Falcone M, Vailati F, Pasticci MB, Perez M, Raglio A, Rumpianesi F, Scuderi C, Suter F, Venditti M, Venturelli C, Ravasio V, Codeluppi M, Stefani S. Changing Italian nosocomial-community trends and heteroresistance in Staphylococcus aureus from bacteremia and endocarditis. Eur J Clin Microbiol Infect Dis. 2012 May;31(5):739-45. doi: 10.1007/s10096-011-1367-y. Epub 2011 Aug 7. PMID 21822974